CLINICAL TRIAL: NCT02956525
Title: Phase I Clinical Study, Open-label, Randomized, Parallel to Evaluate the Safety of the 200 mg Dexibuprofen Following Single and Multiple Dose Oral Administration in Healthy Participants of Both Sexes Under Fasting and Fed Conditions.
Brief Title: Phase I Study to Evaluate the Safety of Dexibuprofen 200mg Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DEXAPS0716OR-LD
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dexibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexibuprofen 200 mg - Fed (Experimental): Fed condition
  Interventions: Drug: Dexibuprofen
- Dexibuprofen 200 mg - Fasting (Experimental): Fasting condition
  Interventions: Drug: Dexibuprofen

INTERVENTIONS:
Drug: Dexibuprofen — Dexibuprofen 200 mg

SUMMARY:
Phase I Study to Evaluate the Safety of Dexibuprofen 200mg (Apsen Pharmaceuticals A / S.) After a Single and Multiple Dose Oral Administration in Healthy Participants of Both Sexes Under Fasting and Fed Conditions.

DETAILED DESCRIPTION:
A single oral dose of test medicine will be administered to participants in a practical period with the aid of 200 mL of water at room temperature. During administration, participants should stay in seated position. Participants will be confined at least 12 hours prior to administration and will remain for about 24 hours after the same, totaling about 36 hours of confinement.

After 36 hours of confinement the participantes will proceed to the multi-dose use phase for seven days in fed conditions.

To assess safety, an evaluation of the vital signs, laboratory tests and health status of the participants will be carried out throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant able to understand and sign the informed consent of the study;
* Healthy research participant, of both sexes, aged between 18 and 50 years, with BMI between 18.50 and 29.99 kg / m2;
* Participant considered healthy by evaluating the medical history, vital signs and general clinical examination;
* The results of clinical laboratory tests (biochemistry, hematology, serology, urinalysis and ECG certified by cardiologists) within the normal range established by the laboratory or changes that are considered not clinically significant by study physician.

Exclusion Criteria:

* History of any major surgery in the last three months;
* History present or previous history of any cardiac event, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric, hematologic, considered by the investigator as clinically significant and can endanger the participant's health;
* History of chronic alcohol abuse, drugs, drugs and / or smoking in the last 6 months;
* Known hypersensitivity to dexibuprofen, ibuprofen or its related (other nonsteroidal anti-inflammatory drugs) as well as components present in the formulation;
* History of use of drugs that potentially interfere with the kinetics / dynamics dexibuprofen or any other medication considered clinically significant by the investigator with time less than 7 times of drug half-life preceding the period of inclusion;
* Regular consumption of grapefruit and / or their derivatives;
* Pregnant women and nursing mothers;
* Donation or loss of 450 ml or more of blood within 3 months before the study and / or hospitalization for any reason, up to 4 weeks before the beginning of it.
* Participation in any clinical trial in the last 12 months preceding the start of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the drug through the incidence and classification of adverse events following single and multiple dose administration. | 40 days
  Adverse events both recorded in the single-dose and multiple-dose

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of the drug dexibuprofen at 200 mg concentration after single dose oral administration under fasting and fed conditions. | 36 hours
  Evaluation of pharmacokinetic parameters: Tmax, Cmax, AUC, DV, Kel, CL and T1/2.

CONTACTS AND LOCATIONS:
Overall Officials: Dra. Regina Mayumi Doi, MD, Principal Investigator — Azidus
Locations (1):
- Azidus laboratories Ltd., Valinhos, São Paulo, Brazil